CLINICAL TRIAL: NCT02912819
Title: Individualized Lung Recruitment Maneuver Guide by Pulse-oximetry in Anesthetized Patients
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: Instituto de Investigacion Sanitaria INCLIVA (Other)
Responsible Party: Principal Investigator, Carlos Ferrando, MD, PhD, Fundación para la Investigación del Hospital Clínico de Valencia
Other Study IDs: SpO2-guide RM
Record Dates: First submitted 2016-09-11; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Abdominal Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Open-lung approach — Increase and decrease in airway pressure to open the lung and keep them opened.

SUMMARY:
General anesthesia and mechanical ventilation promotes atelectasis and airway closure. The open-lung approach (OLA) strategy restores the functional residual capacity. Pulse oximetry hemoglobin saturation (SpO2) using room air can diagnose shunt induced by lung collapse during general anesthesia and the SpO2 breathing air was useful to detect the lung´s opening and closing pressure during a recruitment maneuver (RM) in morbidly obese anesthetized patients.

Investigators hypothesized that the SpO2 breathing air can personalize the open-lung approach.

DETAILED DESCRIPTION:
Increase in airway pressure until the SpO2 reaches 97% (lung´s opening pressure) during the incremental positive end-expiratory (PEEP) limb. Decrease in the PEEP level until the SpO2 decreases bellow 97% (lung´s closing pressure)

ELIGIBILITY:
Inclusion Criteria:

* Non-obese patients with ASA physical status I-III undergoing elective abdominal laparoscopic surgery with an expected operating time of less than 2 hours were included.

Exclusion Criteria:

* age of <18 years,
* preoperative SpO2 ≤97% while breathing room air, and
* patients with previous known cardiac or respiratory disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included all patients with ASA status I-III scheduled for elective abdominal laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
open-lung condition | During the experimental protocol (Intraoperative)
  The role of the SpO2 to detect lung´s closing and opening pressures was evaluated by the discrete receiver operating characteristic (ROC) analysis. With PtpEE and PaO2/FIO2 as the reference methods, a binary classification of "1" to the open-lung condition defined as positive PtpEE or PaO2/FIO2 >400 mmHg and "0" presence of lung collapse defined as negative PtpEE or PaO2/FIO2 <400 mmHg. Also, a value of "1" was assigned when the SpO2 was ≥ 97% and a value of "0" when the value was < 97%.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia and Critical Care; Hospital Clinico Universitario, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Shared data will be anonymous

REFERENCES:
- [Background] Tusman G, Groisman I, Fiolo FE, Scandurra A, Arca JM, Krumrick G, Bohm SH, Sipmann FS. Noninvasive monitoring of lung recruitment maneuvers in morbidly obese patients: the role of pulse oximetry and volumetric capnography. Anesth Analg. 2014 Jan;118(1):137-44. doi: 10.1213/01.ane.0000438350.29240.08. PMID 24356163
- [Background] Ferrando C, Mugarra A, Gutierrez A, Carbonell JA, Garcia M, Soro M, Tusman G, Belda FJ. Setting individualized positive end-expiratory pressure level with a positive end-expiratory pressure decrement trial after a recruitment maneuver improves oxygenation and lung mechanics during one-lung ventilation. Anesth Analg. 2014 Mar;118(3):657-65. doi: 10.1213/ANE.0000000000000105. PMID 24557111